CLINICAL TRIAL: NCT00957853
Title: An Exploratory Study to Assess the Modulation of Biomarkers in Patients With Squamous Cell Carcinomas of the Head and Neck Randomized to Receive Preoperative Treatment With Cetuximab and/or IMC-A12, an Anti-insulin-like Growth Factor-1 Receptor Monoclonal Antibody
Brief Title: Preoperative Treatment With Cetuximab and/or IMC-A12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0342; NCI-2011-03039 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Cancer; Squamous cell carcinoma of the head and neck; HNSCC; Cetuximab; IMC-A12; Tumor; Biomarkers; Phospho-AKT; Surgical resection
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Neoplasms | interventions — Cetuximab; cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Cetuximab (Experimental): Cetuximab: 400 mg/m2 i.v. over 120 minutes on week 1, and 250 mg/m2 on week 2 and 3 i.v. over 60 minutes
  Interventions: Drug: Cetuximab; Procedure: Surgical tumor resection
- Group 2: IMC-A12 (Experimental): IMC-A12: 6 mg/kg/week i.v. over 1 hour on weeks 1 and 2 and 3.
  Interventions: Drug: IMC-A12; Procedure: Surgical tumor resection
- Group 3: Cetuximab + IMC-A12 (Experimental): Cetuximab: 400 mg/m2 i.v. over 120 minutes on week 1, and 250 mg/m2 on week 2 and 3 i.v. over 60 minutes.
  IMC-A12: 6 mg/kg/week i.v. over 1 hour on weeks 1 and 2 and 3.
  Interventions: Drug: Cetuximab; Drug: IMC-A12; Procedure: Surgical tumor resection

INTERVENTIONS:
Drug: Cetuximab — First dose of 400 mg/m^2 by vein on Days 1 and 8 over 2 hours, second dose of 250 mg/m^2 on week 2 and 3 (if applicable) given over 1 hour.
  Other Names: C225; Erbitux; IMC-C225
  Arms: Group 1: Cetuximab; Group 3: Cetuximab + IMC-A12
Drug: IMC-A12 — 6 mg/kg/week by vein on Days 1 and 8 over 1 hour on weeks 1 and 2 and 3 (if applicable).
  Arms: Group 2: IMC-A12; Group 3: Cetuximab + IMC-A12
Procedure: Surgical tumor resection — Surgical tumor resection on Day 10.

SUMMARY:
The goal of this clinical research study is to give cetuximab and/or IMC-A12 before surgery for squamous cell carcinoma of the head and neck, in order to learn if these study drugs may cause changes in biomarkers. Biomarkers are chemical "markers" in the blood and/or tissue that may be related to a reaction to study treatment.

The safety of the study treatments will also be studied.

DETAILED DESCRIPTION:
The Study Drugs Cetuximab and IMC-A12 are both designed to block proteins that are thought to cause cancer cells to grow. This may help to slow the growth of tumors.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups. There is an equal chance of being assigned to any group.

* Group 1 will receive cetuximab alone.
* Group 2 will receive IMC-A12 alone.
* Group 3 will receive cetuximab and IMC-A12 in combination.

If you are assigned to group 2 or 3 you will have a hearing test within 90 days before starting treatment with the study drug.

Study Treatment:

Groups 1 and 3:

Cetuximab will be given by vein on Days 1 and 8. The first dose will be given over 2 hours. The second dose will be given over 1 hour.

To lower the risk of allergic reaction, Groups 1 and 3 will also receive diphenhydramine by mouth or by vein before the first dose of cetuximab. If the study doctor decides it is needed, diphenhydramine may also be given before the second dose of cetuximab (and the third, if applicable).

Groups 2 and 3:

IMC-A12 will be given by vein over 1 hour on Days 1 and 8.

All Groups:

You will have surgery on Day 10. If for some reason the surgery is delayed, the study doctor may decide that you will receive a third dose of your assigned study drug(s) on Day 15. In that case, cetuximab will be given over 1 hour and/or IMC-A12 will be given over 1 hour, depending on which group you are in.

You will sign a separate consent form that describes the surgery and its risks in more detail.

Study Tests:

Within 5 days before your second dose of study drug(s), and again within 5 days before your third dose (if applicable), the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will be asked about any side effects you may be experiencing.
* You will have a physical exam, including measurement of vital signs.
* Blood (about 3 teaspoons) will be drawn for routine tests.

On the day before surgery, you will have a CT scan or MRI of the head and neck. If needed, these tests can instead be done before surgery but sometime after the last dose of the study drug(s).

On the day of surgery, blood (about 3 teaspoons) will be drawn for routine tests and your vital signs will be measured. If needed, these tests can instead be done up to 2 days before surgery.

Length of Study Drug Dosing:

After your last dose of the study drug(s), on Day 8 or Day 15, your participation in the study treatment period will be over. You will be taken off the study drug(s) early if the disease gets worse or intolerable side effects occur.

Follow-Up:

If you return to the clinic within 30 days after surgery, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any side effects that may have occurred.

Otherwise if you do not have a visit scheduled during that time, the study staff will call you by phone instead. You will be asked how you are doing.

If you are experiencing side effects from the study drug(s) at the time of the follow-up visit or call, you may have additional follow-up if the doctor decides it is needed. The follow-up tests, procedures, and schedule will be the doctor's decision depending on the side effects.

You will have a repeat hearing test within 90 days after surgery if you received at least 1 dose of IMC-A12.

Long-Term Follow-Up:

On a long-time basis after surgery, the study staff may review your medical record to collect information about your health. During this time, you or your family members may be contacted and asked to confirm or provide information about your health. The contact may occur during clinic visits or by phone, mail, or e-mail.

This is an investigational study. Cetuximab is commercially available and FDA approved to treat squamous cell carcinoma that has spread or come back, in patients who did not respond to platinum-based therapy.

Using cetuximab in combination with surgery is investigational.

IMC-A12 is not FDA approved or commercially available. At this time, IMC-A12 is only being used in research.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-confirmed diagnosis of squamous cell carcinoma of the head and neck (excluding carcinomas of the nasopharynx types II and III according to the World Health Organization criteria), for whom surgical resection of the tumor is planned as part of the treatment. Patients with skin squamous cell carcinomas of the head and neck region will also be included in this study.
2. There is availability of a baseline, paraffin-embedded, tumor specimen for biomarker evaluation. No anti-neoplastic treatment is allowed between the time from obtaining the baseline tumor specimen and randomization. If a baseline tumor specimen is not available, a biopsy of the tumor will be performed prior to randomization.
3. Prior treatment with biological agents targeted to the epidermal growth factor receptor is allowed, provided the time from last exposure to this treatment was >/= 6 months.
4. The patient has a fasting serum glucose < 130 mg/dL and HbA1C < 7.0%. Patients with a history of diabetes mellitus are allowed to participate, provided that they are on a stable dietary or therapeutic regimen for this condition.
5. The patient has adequate renal function, defined by serum creatinine </= 1.5 x the institutional upper limit of normal (ULN), or creatinine clearance >/=60 mL/min for patients with creatinine levels above the ULN.
6. Because the teratogenicity of cetuximab and IMC-A12 is not known, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
7. The patient is age >/= 18 years.
8. The patient or the patient's legally authorized representative has the ability to understand and the willingness to sign a written informed consent document.
9. ECOG performance status of 0-2.

Exclusion Criteria:

1. Patients receiving any other agent (investigational or not) with potential anti-neoplastic activity within 3 weeks prior to obtaining the baseline tumor specimen for biomarker evaluation.
2. Patients receiving concomitant radiation.
3. Prior treatment with an agent targeted at the insulin-like growth factor-1 receptor.
4. History of allergic reactions attributed to compounds of chemical and biological composition similar to those of cetuximab or IMC-A12.
5. Pregnant patients, or patients who are breast feeding (patients who have a positive pregnancy test within the first 30 days before the first dose of treatment are excluded).
6. Patients with uncontrolled illnesses which, in the opinion of the investigator, could be aggravated by the administration of the study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-10-17 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maura Gillison, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 16 patients were enrolled in the study; however only 15 patients were started on the trial since 1 subject withdrew consent for the study.
Groups:
- Cetuximab: Subjects received Cetuximab at 400 mg/m2 loading dose and 250 mg/m2 subsequently for 1-2 doses
- IMC-A12: Subjects received IMC-A12 at 6 mg/kg
- Cetuximab + IMC-A12: Subjects received Cetuximab at 400 mg/m2 loading dose and 250 mg/m2 subsequently for 1-2 doses. Subjects received IMC-A12 at 6 mg/kg
Period: Overall Study
Arm/Group | Cetuximab | IMC-A12 | Cetuximab + IMC-A12
Started | 4 | 6 | 5
Randomization | 4 | 6 | 5
Neoadjuvant Tx Completion | 3 | 6 | 5
Completed | 3 | 6 | 5
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab | IMC-A12 | Cetuximab + IMC-A12 | Total
Number analyzed (Participants) | 4 | 6 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 2 | 4 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 3 | 4 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 5 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: AKT Modulation
Description: An IHC scoring system used to quantify phospho-Akt levels based on staining intensity x extension. Staining intensity graded as undetectable (0), weak (1), medium (2), or strong (3). Staining extension graded as percentage of positive cells per high power field at x20 magnification. Final score will therefore range from 0 to 300. Modulation of phospho-Akt (difference in IHC score between the surgical specimen and the baseline biopsy) and other biomarkers compared between any two of the three treatment arms with the use of the Wilcoxon rank sum test. Type I error of alpha=0.05 (two-sided test) used. Correlation between biomarkers and molecular response or toxicity performed in an exploratory fashion.
Time Frame: Biopsy at baseline and surgery (surgery should be within 10 days of last treatment)
Population: Due to early termination of the study, data could not be collected for this outcome.
Arm/Group | Cetuximab | IMC-A12 | Cetuximab + IMC-A12
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response to treatment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 4 months post treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab | IMC-A12 | Cetuximab + IMC-A12
Number analyzed (Participants) | 4 | 6 | 5
Participants
  Stable Disease/No Change | 3 | 4 | 5
  Progressive Disease | 0 | 2 | 0
  Inevaluable | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Mortality and SAE's were assessed from the first dose of study treatment to 30 days following the last dose of drug.
Description: Adverse events were assessed according to the CTCAE
Arm/Group | Cetuximab | IMC-A12 | Cetuximab + IMC-A12
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/4 | 2/6 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=4) | IMC-A12 (N=6) | Cetuximab + IMC-A12 (N=5)
Acneiform rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Fever without Neutropenia (General disorders) | 0 | 0 | 1
Hot flashes (General disorders) | 0 | 1 | 0
Mucositis-symptomatic (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Pain(headache) (General disorders) | 2 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rigors/Chills (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT00957853/Prot_SAP_000.pdf